CLINICAL TRIAL: NCT04957173
Title: Intervention Intensive Sur le Mode de Vie Chez Les Patients Atteints d'obésité Avec un diabète de Type 2 avancé Insuline-traité : un Projet Pilote
Brief Title: Intensive Lifestyle Intervention in Patients With Insulin-treated Type 2 Diabetes: a Pilot Project
Acronym: ILIAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was difficult, and the investigator decided to close the study.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILIAD-CHUM
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive lifestyle intervention (Other): Participants will undergo an intensive lifestyle intervention, implemented virtually by a medical team with expertise in the management of T2DM. This team will be made up of an endocrinologist, a nutritionist and a nurse.
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — The intervention includes a total of 17 virtual meetings and aims to achieve a weight loss of 0.8 to 1% of the initial weight per week.
  This will include 3 successive phases:
  1. A significant calorie restriction (A minimum deficit of 800 kcal / day of their daily energy expenditure) for a period of 4 weeks;
  2. A moderate calorie restriction (minimum deficit of 500 kcal / day of their daily energy expenditure) for a period of 4 weeks;
  3. A maintenance phase of weight loss for 16 weeks.
  4. An optional phase of monthly follow-ups for a period of 3 months (no intervention)

SUMMARY:
This study is a pilot study carried out to assess the feasibility, safety and effectiveness of an intensive lifestyle intervention, implemented virtually by a multidisciplinary team, in patients living with advanced insulin-treated T2DM. This 24-week study will include 2 pre-intervention virtual visits and 15 virtual visits during the intervention.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2DM) has increased rapidly over the past decades. This chronic condition, strongly associated with abdominal obesity, leads to serious complications. Traditional recommendations for the management of T2DM mainly suggest the use of drugs to control blood sugar and the concomitant risk factors. However, this approach can be expensive and some therapies have significant side effects. Although programs aimed at improving lifestyle habits are essential in the management of T2DM, the implementation of these programs involves many challenges such as the need for patients to travel and access to a multidisciplinary team.

A few studies have recently proposed that one can induce remission of T2DM. Considering that this disease appears to be the result of metabolic stress induced by an excessive accumulation of fat in the internal organs, the reduction of this excess of lipids by a significant weight loss could reduce the metabolic stress and modify the progression of the disease. disease.

The implementation of a virtual lifestyle intervention could make it possible to follow up patients who do not have access to a multidisciplinary team nearby or who are unable to travel.

The objective of this project is to assess the feasibility of the nutritional intervention by measuring food intake, eating behaviors and factors facilitating or limiting adherence to the intervention. As well as to examine the effect of this intervention on weight loss and waist circumference; doses of insulin and other drugs to treat T2DM, dyslipidemia and high blood pressure; glycemic control and possible complications; eating behaviors and quality of life.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 75, BMI 27 to 45 kg / m2
2. Diagnosed T2DM
3. Insulin-treated for a minimum of 5 years
4. Having a glycated hemoglobin <9.5% (HbA1c dating ≤3 months)
5. Having internet and telephone access to enable monitoring of the intervention and remote blood glucose monitoring
6. If treated with a glucagon like peptide-1 (GLP-1), must be on a stable dose for a minimum of 6 months
7. Having good autonomy in managing medication (including insulin) and preparing meals.

Exclusion criteria:

1. A diagnosis of T2DM with a tendency to ketosis
2. A history of ketoacidosis associated with taking an SGLT2 inhibitor
3. Medical history of eating disorders
4. Severe hypoglycemia in the past year or decreased perception of hypoglycemia determined by Clarke's method with a score ≥ 4 (17)
5. A history of gastrointestinal tract surgery that alters the ability to absorb nutrients (weight loss surgery, short bowel, etc.) [cholecystectomy or appendectomy are not exclusion criteria]
6. A history of pancreatic insufficiency, advanced liver disease or liver transplant [Hepatic steatosis is not an exclusion criterion]
7. Active cancer under treatment or a history of cancer with active treatment in the past year (basal cell carcinoma is not an exclusion criteria)
8. Daily fluid restriction
9. A pregnant / breastfeeding participant, wishing to be pregnant during the study period or having given birth less than one year before the start of the study
10. The presence of advanced complications of T2DM (renal failure with estimated glomerular filtration rate <30 ml / min / 1.73m2, proliferative diabetic retinopathy, severe neuropathy)
11. Drug or alcohol use in the past 12 months. Defined by more than 2 drinks per day or more 10 per week for women, and more than 3 drinks per day or more than 15 per week for men.
12. Advanced fragility (See the score which is in the recommendations of Diabetes Canada chapter elderly people)
13. A macrovascular episode (heart attack, stenting, coronary bypass surgery or stroke less than 6 months ago.
14. An active wound Additional to the inclusion/exclusion criterias, the PI will determine the inclusion of the participant to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be weight loss in the participants. | 24 weeks
  Weeks 1 to 4: Target weight loss of 1% per week (on average) Weeks 5 to 8: Loss of 0.5% of target weight per week (on average) Weeks 9 to 24: Maintaining target weight